CLINICAL TRIAL: NCT03407365
Title: Clinical Efficacy of A Home-Based Functional Exercise Program in Patients With Patellar Femoral Syndrome Over a 10-Week Period
Brief Title: Home-Based Functional Exercise Program in Patients With Patellar Femoral Syndrome Over a 10-Week Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12-00210
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Patellar Femoral Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Exercises (Experimental): Patients will be given a set of home exercises to perform as part of their rehabilitation home exercise program. They will be initially trained by a research team member and will be given a DVD home exercise video with instructions on how to perform the exercises.
  Interventions: Behavioral: 10 Week Exercise Program
- DVD Program (Active Comparator): Weeks 1-10, subjects will not be prescribed exercise at home. If the DVD program shows to help participants in Group 1, the program and DVD will be provided to Group 2 participants
  Interventions: Behavioral: DVD Program After 10 Weeks

INTERVENTIONS:
Behavioral: 10 Week Exercise Program — Subjects will complete a 10 week exercise program using DVD with instructions provided. Participants will have to do one session of exercise on 5 different days each week for a total of 5 sessions per week, for 10 weeks.
  Arms: Home Exercises
Behavioral: DVD Program After 10 Weeks — If the DVD program shows to help participants in Group 1, the program and DVD will be provided to Group 2 participants
  Arms: DVD Program

SUMMARY:
The purpose of this study is to determine if a 10 week exercise rehabilitation program decreases anterior knee oain (PFPS) and improves function in patients with patellofemoral pain syndrome (PFPS). Individuals (age 18-50) with PFPS will be recruited to participate in this study to see if a 10 week exercise program focusing in core and hip strengthening, lower extremity strengthening foot intrinsic strengthening can decrease pain and increase function.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is a very prevalent condition that presents in great number to patients in physician's offices and has a high recurrence rate. Physical therapy and exercise therapy to strengthen the quadriceps is often prescribed, however recurrence is common. It is hypothesized that PFPS patients have core weakness, hip strength abnormalities and neuromuscular control deficits.

ELIGIBILITY:
Inclusion Criteria:

* Individuals wishing to participate in study voluntarily
* Subjects diagnosed with patella-femoral syndrome. We will ascertain this by asking a few questions, which will not be recorded as they have not been enrolled in the study yet.
* Capable of following and completing a 10 week home exercise program

Exclusion Criteria:

* Individuals with prior knee surgery, tibial plateau fractures, known diagnosis of knee injuries such as meniscus or ligaments tears.
* Individuals unable to participate, i.e. cognitive deficits, weakness or functional deficits to upper extremities.
* Individuals unable to tolerate exercise program

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Kujala Scale for Anterior Knee Pain | 10 Weeks
  13 item knee specific self report questionnaire that documents response to six activities thought to be associated specifically with anterior knee pain syndrome (walking, running, jumping, climbing stairs, squatting and sitting for prolonged periods with knees bent, as well as symptoms such as limp, inability to weight bear through affected the affected limb, swelling, abnormal patellar movement, muscle atrophy and limitation of knee flexion. The maximum score is 100 and lower scores indicate greater pain/disability.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Stokes, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States